CLINICAL TRIAL: NCT01441687
Title: Comparing the Reliability of Expressed Prostatic Secretion (EPS) and Post Massage Urine (PMU) for the Prediction of Prostate Cancer Biopsy Outcome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 08239; NCI-2017-00089 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-09-23; First posted 2011-09-28 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Conditions Influencing Health Status; Healthy; Prostate Cancer
Keywords: Health status unknown; healthy,no evidence of disease
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (PMU) (Experimental): Patients receive digital rectal palpation and then void a spontaneous urine sample for PMU analysis. Patients then undergo a prostate biopsy.
  Interventions: Other: laboratory biomarker analysis; Procedure: transrectal prostate biopsy
- Arm II (EPS) (Experimental): Patients receive DRE with prostatic massage for 30-60 seconds and are then milked at the urethra to provide a collection of EPS. Patients then undergo a prostate biopsy.
  Interventions: Other: laboratory biomarker analysis; Procedure: transrectal prostate biopsy

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies
Procedure: transrectal prostate biopsy — Undergo prostate biopsy

SUMMARY:
This randomized pilot phase I trial studies the best way, either expressed prostatic secretion (EPS) or post massage urine (PMU) biomarkers, of predicting biopsy results in patients undergoing prostate biopsy. Studying samples of urine in the laboratory may help doctors detect prostate cancer. It is not yet known whether EPS or PMU biomarkers are more effective in predicting prostate biopsy results

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine which non-invasive test for prostate cancer, EPS or PMU, is a better predictor of prostate cancer biopsy result. (Part I)

II. To determine whether standardized testing for transmembrane protease, serine 2 (TMPRSS2):ERG Types III and VI is superior to testing for TMPRSS2:ERG Type III in predicting prostate biopsy outcome. (Part I)

III. To expand the sample size utilizing the best TMPRSS2:ERG test and the best specimen type as determined in objective I and II in order to estimate with reasonable accuracy the positive predictive value (PPV) and negative predictive value (NPV) for each test. (Part II)

IV. To expand the biomarker set, to include Prostate Cancer Antigen 3 (PCA3)-ribonucleic acid (RNA), d-glyceraldehyde-3-phosphate dehydrogenase (GADPH)-RNA, prostate-specific antigen (PSA)-RNA, and deoxyribonucleic acid (DNA) methylation levels at glutathione s-transferase pi (GSTP1), adenomatous polyposis coli (APC), retinoic acid receptor beta (RARB), Mitochondrial DNA (MT-DNA) Deletions and ras association (RalGDS/AF-6) domain family 1 (RASSF1), so as to develop an extensive data set for use in multivariate analysis. (Part II)

V. Use multivariate analysis to determine which combination of molecular markers offers the greatest improvements in our ability to predict biopsy outcome over current baseline predictors (Serum PSA and digital rectal examination [DRE]). (Part II)

VI. Estimate PPV and NPVs from this analysis and compare them to the standard assay's performance. (Part II)

OUTLINE: Patients are randomized to 1 of 2 treatment arms. ARM I: Patients receive digital rectal palpation and then void a spontaneous urine sample for PMU analysis. Patients then undergo a prostate biopsy.

ARM II: Patients receive DRE with prostatic massage for 30-60 seconds and are then milked at the urethra to provide a collection of EPS. Patients then undergo a prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* All men who will be undergoing transrectal ultrasound of the prostate (TRUSP) with biopsy in the department of Urology or participating urology clinics for the evaluation of prostate cancer

Exclusion Criteria:

* Men with a previous diagnosis of prostate cancer
* Men without a prior diagnosis of prostate cancer but who have previously undergone a biopsy for a suspicious DRE or PSA
* Men with a prior diagnosis of cancer < 5 years ago, excluding basal cell carcinoma and/or squamous cell carcinoma

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2009-07-14 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2026-02-09 (Estimated)

PRIMARY OUTCOMES:
Determine whether EPS or PMU is a better predictor of prostate cancer biopsy results by measuring and comparing the number of prostatic cells collected | 1 month after sample collection
  Compare assay results in 300 EPS specimens with those from 300 PMU specimens. The gold standard for assay validity is the biopsy result.
Comparison of the area under the curve (AUC) for sensitivity and specificity of TMPRSS2:ERG single and double fusion assays and biopsy results in patients with prostate cancer, undergoing prostate screening | 1 month after sample collection
  Perform TMPRSS2:ERG type III and TMPRSS2:ERG type IV assays on each specimen. The gold standard for assay validity is the biopsy result.

SECONDARY OUTCOMES:
Comparison of the AUC for sensitivity and specificity of the methylation status of the androgen receptor (AR) and GSTP1 promoter, APC and RARB and biopsy results in men with prostate cancer, undergoing prostate screening | 1 month after sample collection
  The gold standard for assay validity is the biopsy result.
Determine by comparison of AUCs which combination of molecular markers offers the greatest improvements in our ability to predict biopsy outcome over current baseline predictors (serum PSA and DRE) | 1 month after sample collection
  The gold standard for assay validity is the biopsy result.
Comparison through the AUCs of the association of EPS or PMU TMPRSS2:ERG fusion assay and methylation of the GSTP1 promoter, APC, RARB assays and PCA3 to the results of TRUSP and biopsy in men with unknown prostate cancer status | 1 month after sample collection
  The gold standard for assay validity is the biopsy result.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Smith, PhD, Principal Investigator — City of Hope Medical Center
Locations (5):
- United States (5):
  - Chinn & Chinn Urology Associates, Inc., Arcadia, California
  - City of Hope Medical Center, Duarte, California
  - Citrus Valley Urologic Medical Group, Glendora, California
  - Dr. Felix Chi-Ming Yip, Monterey Park, California
  - City of Hope- South Pasadena Cancer Center, South Pasadena, California